CLINICAL TRIAL: NCT06508476
Title: The Efficacy of Amnion Chorion Allograft in Management of Type 1 Gingival Recession. (Randomized Clinical Trial)
Brief Title: The Efficacy of Amnion Chorion Allograft in Management of Gingival Recession.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina gerges, Principal investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 857
Record Dates: First submitted 2024-07-03; First posted 2024-07-18 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2024-07

CONDITIONS: Gingival Recession, Localized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: two groups Group 1 contains 16 patients and will be treated by CAF and SCTG. Group 2 also contains 16 patients and will be treated by CAF and ACM (bioxclude, snoasis medical, Denver, Co.USA).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Amnion chorion allograft (Experimental): participants will receive amnion chorion with coronally advanced flap
  Interventions: Biological: Amnion Chorion membrane
- Connective tissue graft (Active Comparator): participants will receive connective tissue graft with coronally advanced flap
  Interventions: Procedure: connective tissue graft

INTERVENTIONS:
Biological: Amnion Chorion membrane — it is a placental allograft.
  Arms: Amnion chorion allograft
Procedure: connective tissue graft — it is an autograft
  Arms: Connective tissue graft

SUMMARY:
the main goal of this clinical trial is to test the efficacy of amnion Chorion allograft in managing gingival recession. The main questions it aims to answer are: Is it effective in treating gingival recession, and how it compares to connective tissue graft.

DETAILED DESCRIPTION:
Gingival recession (GR) is characterized by apical migration of soft tissue margin beyond the cemento-enamel junction (CEJ) or the platform of an implant.

Gingival recession is a common daily finding in every practice. As patients are more concerned with a pleasing smile, root exposure is a growing concern . Moreover, discomfort and inability to perform oral hygiene result from exposed root hypersensitivity. It affects the patient's abilities to maintain adequate plaque control which eventually complicates the situation more. It is advisable to augment tissues and increase keratinized tissue (KT) band to reduce discomfort and obtain an aesthetic smile.

multiple treatment modalities are available for treating gingival recession such as Pedicle flaps (coronally advanced flap (CAF), semilunar flap, laterally sliding flap (lSD), and double papilla flap), Free gingival graft (FGG), Subepithelial connective tissue graft (SCTG), Guided tissue regeneration. Modified coronally advanced tunnel, Vestibular incision subperiosteal tunnel access (VISTA), Pinhole technique (PST).

Size and number of recession defects, KT band, interproximal attachment level, depth vestibule and frenum pull are among factors to determine which procedure is suitable for that type of recession.

For single-type recession (localized or isolated), the use of CAF with SCTG is favorable for both root coverage and KT gain. According to the American Academy of Periodontology regeneration workshop "for Miller class 1 and 2 single-tooth recession defects, SCTG procedures provide the best outcome ". Using CAF combined with SCTG is considered the gold standard treatment for localized recession defects. SCTG improves root coverage, KT gain, and clinical attachment levels. Using SCTG helps stabilize CAF, increase root coverage predictability, and increase soft tissue thickness. CAF with SCTG is a predictable technique to increase root coverage, decrease recession depth, and increase KT width and thickness.

However, obtaining an SCTG has some drawbacks such as the need for a second surgical site to harvest graft increases treatment time and patient morbidity. Bleeding and postoperative discomfort are common after graft harvesting. Another issue is a limited amount of tissue is also a concern in multiple defect cases. Patients' willingness to retreat was affected by previous autogenous grafting.

Recently, the use of placental membranes is introduced as a suitable substitute for SCTG. The human placenta is composed of two membranes inner amniotic and outer chorionic membranes. These membranes secrete anti-inflammatory cytokines and growth factors such as platelet-derived growth factor AA (PDGF-AA) and vascular endothelial growth factor (VEGF). These membranes have anti-inflammatory, angiogenic, antifibrotic, and antimicrobial effects. Furthermore, they have low immunogenicity and improve epithelization. They have been widely used in medicine since the 1910s with increasing clinical applications from wound care and ophthalmology, to plastic surgery.

There is a growing interest in using placental allografts as a substitute for conventional membranes in oral surgical procedures. They are used for root coverage as a substitute for SCTG as these membranes contain different types of collagen, proteoglycans, laminin, and bioactive factors which help in binding gingival epithelial cells to the root surface. They act as reservoirs of stem cells which promote cell differentiation, stimulate healing, and help in revascularization.

So in this study, it is proposed to evaluate Amnion Chorion membrane in the management of gingival recession type 1 in comparison to SCTG.

Aim of the study The primary outcome is to evaluate the effectiveness of the Amnion Chorion membrane (ACM) in the management of gingival recession type 1 (RT1).

The secondary outcome is to compare between ACM and subepithelial connective tissue graft in the treatment of recession defect type 1 (RT1).

ELIGIBILITY:
Inclusion Criteria:

1. Selected patients of both sexes are 25-45 years old.
2. Patients are systemically healthy based on the questionnaire dental modification of the Cornell index.
3. O'Leary index (1972) is less than 10% (the surgical therapy is not initiated until the patient reaches the 10% level or less of plaque accumulation).
4. Buccal recession defects are classified RT1 according to Cairo's classification (2011).
5. Clinical indication and/or patient request for recession coverage.

Exclusion Criteria:

1. RT2 and RT3 recession defects.
2. Pregnant female.
3. Smokers.
4. Patients with special needs or with any mental problems.
5. All patients are using any kind of medication that could interfere with the healing of periodontal tissues. Such as chemotherapy and radiotherapy.
6. Teeth with root carious lesions.
7. Rotated and extruded teeth.
8. Patients underwent any prior periodontal surgery in the relevant region.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-22 (Actual)

PRIMARY OUTCOMES:
recession depth | changes in millimeters from base line to follow up after 6 months
  recession depth is measured from CEJ to the gingival margin in millimeters.

SECONDARY OUTCOMES:
Recession Width | changes in millimeters from base line to follow up after 6 months
  it is measured at the widest point from the mesial gingival margin to the distal gingival margin in millimeters
the height of keratinized gingiva | changes in millimeters from base line to follow up after 6 months
  it is measured in millimeters as the distance from the mucogingival junction to the gingival margin, with the mucogingival junction location determined using a visual method.
Probing pocket depth | changes in millimeters from base line to follow up after 6 months
  it is measured as the distance from the gingival margin to base of pocket.
percentage of root coverage | changes in percentile from base line to follow up after 6 months
  it will be calculated as [pre-operative gingival recession depth - post-operative recession depth]/ [preoperative recession depth] * 100%

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Khalil, professor, Study Chair — Minia University; Aya Mohammed, Lecturer, Study Director — Minia University
Locations (1):
- faculty of dentistry, Minia University, Minya, Other, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Data are available indefinitely at (Link to be included).

REFERENCES:
- [Background] Amine K, El Amrani Y, Chemlali S, Kissa J. Alternatives to connective tissue graft in the treatment of localized gingival recessions: A systematic review. J Stomatol Oral Maxillofac Surg. 2018 Feb;119(1):25-32. doi: 10.1016/j.jormas.2017.09.005. Epub 2017 Sep 9. PMID 28893718
- [Background] Cairo F, Nieri M, Cincinelli S, Mervelt J, Pagliaro U. The interproximal clinical attachment level to classify gingival recessions and predict root coverage outcomes: an explorative and reliability study. J Clin Periodontol. 2011 Jul;38(7):661-6. doi: 10.1111/j.1600-051X.2011.01732.x. Epub 2011 Apr 20. PMID 21507033
- [Background] Chambrone L, Chambrone D, Pustiglioni FE, Chambrone LA, Lima LA. Can subepithelial connective tissue grafts be considered the gold standard procedure in the treatment of Miller Class I and II recession-type defects? J Dent. 2008 Sep;36(9):659-71. doi: 10.1016/j.jdent.2008.05.007. Epub 2008 Jun 26. PMID 18584934
- [Background] Chambrone L, Pannuti CM, Tu YK, Chambrone LA. Evidence-based periodontal plastic surgery. II. An individual data meta-analysis for evaluating factors in achieving complete root coverage. J Periodontol. 2012 Apr;83(4):477-90. doi: 10.1902/jop.2011.110382. Epub 2011 Aug 22. PMID 21859324
- [Background] Chambrone L, Salinas Ortega MA, Sukekava F, Rotundo R, Kalemaj Z, Buti J, Pini Prato GP. Root coverage procedures for treating localised and multiple recession-type defects. Cochrane Database Syst Rev. 2018 Oct 2;10(10):CD007161. doi: 10.1002/14651858.CD007161.pub3. PMID 30277568
- [Background] Chambrone L, Tatakis DN. Periodontal soft tissue root coverage procedures: a systematic review from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S8-51. doi: 10.1902/jop.2015.130674. PMID 25644302
- [Background] de Sanctis M, Zucchelli G. Coronally advanced flap: a modified surgical approach for isolated recession-type defects: three-year results. J Clin Periodontol. 2007 Mar;34(3):262-8. doi: 10.1111/j.1600-051X.2006.01039.x. PMID 17309597
- [Background] Gulameabasse S, Gindraux F, Catros S, Fricain JC, Fenelon M. Chorion and amnion/chorion membranes in oral and periodontal surgery: A systematic review. J Biomed Mater Res B Appl Biomater. 2021 Aug;109(8):1216-1229. doi: 10.1002/jbm.b.34783. Epub 2020 Dec 22. PMID 33354857
- [Background] Imber JC, Kasaj A. Treatment of Gingival Recession: When and How? Int Dent J. 2021 Jun;71(3):178-187. doi: 10.1111/idj.12617. Epub 2021 Jan 29. PMID 34024328
- [Background] Madeley E, Duane B. Coronally advanced flap combined with connective tissue graft; treatment of choice for root coverage following recession? Evid Based Dent. 2017 Mar;18(1):6-7. doi: 10.1038/sj.ebd.6401215. PMID 28338039
- [Background] Maity S, Priyadharshini V. Comparison of chorion allograft and subepithelial connective tissue autograft in the treatment of gingival recession- A randomized controlled clinical trial. J Oral Biol Craniofac Res. 2023 Mar-Apr;13(2):104-110. doi: 10.1016/j.jobcr.2022.12.002. Epub 2022 Dec 5. PMID 36578557
- [Background] Moraschini V, Barboza Edos S. Use of Platelet-Rich Fibrin Membrane in the Treatment of Gingival Recession: A Systematic Review and Meta-Analysis. J Periodontol. 2016 Mar;87(3):281-90. doi: 10.1902/jop.2015.150420. Epub 2015 Nov 12. PMID 26561997
- [Background] Moraschini V, Calasans-Maia MD, Dias AT, de Carvalho Formiga M, Sartoretto SC, Sculean A, Shibli JA. Effectiveness of connective tissue graft substitutes for the treatment of gingival recessions compared with coronally advanced flap: a network meta-analysis. Clin Oral Investig. 2020 Oct;24(10):3395-3406. doi: 10.1007/s00784-020-03547-3. Epub 2020 Aug 26. PMID 32851531
- [Background] Mounssif I, Stefanini M, Mazzotti C, Marzadori M, Sangiorgi M, Zucchelli G. Esthetic evaluation and patient-centered outcomes in root-coverage procedures. Periodontol 2000. 2018 Jun;77(1):19-53. doi: 10.1111/prd.12216. Epub 2018 Mar 4. PMID 29504166
- [Background] Pini-Prato G. The Miller classification of gingival recession: limits and drawbacks. J Clin Periodontol. 2011 Mar;38(3):243-5. doi: 10.1111/j.1600-051X.2010.01655.x. Epub 2010 Dec 15. No abstract available. PMID 21158897
- [Background] Stefanini M, Marzadori M, Aroca S, Felice P, Sangiorgi M, Zucchelli G. Decision making in root-coverage procedures for the esthetic outcome. Periodontol 2000. 2018 Jun;77(1):54-64. doi: 10.1111/prd.12205. Epub 2018 Mar 4. PMID 29504173
- [Background] Tavelli L, Barootchi S, Di Gianfilippo R, Kneifati A, Majzoub J, Stefanini M, Zucchelli G, Wang HL. Patient experience of autogenous soft tissue grafting has an implication for future treatment: A 10- to 15-year cross-sectional study. J Periodontol. 2021 May;92(5):637-647. doi: 10.1002/JPER.20-0350. Epub 2020 Oct 3. PMID 32946124